CLINICAL TRIAL: NCT06970795
Title: An Open-lable, Multicenter Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Efficacy of SYS6040 for Injection as a Single Agent in Participants With Advanced Solid Tumors
Brief Title: A Study of SYS6040 for Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS6040
Record Dates: First submitted 2025-04-02; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer; Other Advanced Solid Tumors
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Injections

STUDY DESIGN:
Intervention Model Description: This study is the first-in-human Phase I study of SYS6040 for injection, comprising two phases: Dose escalation with backfill (Phase Ia) and cohort expansion (Phase Ib).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYS6040 for injection as single agent (Experimental)
  Interventions: Drug: SYS6040 for injection

INTERVENTIONS:
Drug: SYS6040 for injection — Intravenous infusion; including dose escalation and backfilling (5 preset dose groups) and cohort expansion.
  Treatment Period: All subjects receive trial treatment until disease progression, death, intolerance of toxicity, loss to follow-up, withdrawal of consent, or end of the trial (whichever occurs first)

SUMMARY:
This study is the first-in-human Phase I study of SYS6040 for injection, comprising two phases: Dose escalation with backfill (Phase Ia) and cohort expansion (Phase Ib).The planned study population consists of subjects with advanced solid tumors.The objective is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of SYS6040 for injection as monotherapy in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The dose escalation phase utilizes a BOIN design for dose escalation. Subjects in five predefined dose groups will administer investigational product via intravenous infusion. Subjects will be enrolled in groups of 3 for treatment.The first treatment cycle (21 days) will serve as the DLT observation window, with dose escalation/de-escalation decisions based on DLT occurrences.

Each cohort is planned to enroll 20-40 subjects, receiving RP2D doses every 3 weeks (Day 1).

Subjects will receive RP2D doses in 21-day treatment cycles until PD, intolerable toxicity, consent withdrawal, loss to follow-up, investigator-determined unsuitability for continued treatment, death, or study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1）Aged ≥18 years; 2) Subjects with histologically or cytologically confirmed advanced solid tumors who have failed standard therapy, are intolerant to standard therapy, or have no options of standard of care. During cohort expansion, subjects will be enrolled as follows: Cohort 1: SCLC subjects who failed or were intolerant to at least one prior platinum-containing chemotherapy regimen; Cohort 2: Subjects with DLL3-positive malignant solid tumors who failed standard therapy, are intolerant to standard therapy, or have no options of standard of care.

3) At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST v1.1); 4) ECOG score of 0 or 1; 5) Life expectancy ≥3 months; 6) Laboratory parameters meeting the following criteria:

1. Neutrophil count ≥1.5×109/L;
2. Platelet count ≥100×109/L;
3. Hemoglobin ≥9 g/dL;
4. Total bilirubin ≤1.5×ULN, ALT and AST ≤2.5×ULN (In cases with liver metastases: total bilirubin ≤3×ULN and ALT/AST ≤5×ULN);
5. Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min;
6. International Standardized Ratio (INR) or activated partial thromboplastin time (APTT) ≤1.5×ULN.

a. Fertile males and females must use reliable contraception throughout the study period and for 9 months after the last dose. Females aged 18-60 years must have negative blood pregnancy results within 7 days before the first dose.

7) Understand and voluntarily sign the informed consent form (ICF).

Exclusion Criteria:

1. Having received systemic antitumor therapy within 4 weeks before first dose, including: Chemotherapy, macromolecular targeted therapy, antiangiogenic therapy, biotherapy, immunotherapy, radiotherapy (except palliative radiotherapy for bone metastasis pain relief), except:

   1. Oral fluorouracil agents and small molecule targeted drugs within 2 weeks before first dose or within 5 half-lives (whichever is longer);
   2. Traditional Chinese medicines with antitumor indications within 2 weeks before first dose.
2. Used or required to use strong CYP3A4 inhibitors/inducers within 2 weeks before first dose or during the study;
3. Previous treatment with antibody-drug conjugates (ADCs) containing topoisomerase I inhibitors as payload;
4. Having received systemic corticosteroid therapy (>10 mg prednisone equivalent daily for >7 days) or other immunosuppressants within 2 weeks before treatment initiation (inhaled/topical steroids or adrenal replacement therapy >10 mg prednisone equivalent permitted without active autoimmune disease);
5. Having received transfusion, EPO, TPO, IL-11, G-CSF or GM-CSF therapy within 2 weeks before first dose;
6. Having used or required to use QT-prolonging/shortening drugs within 7 days before first dose or during C-QTc study period, or have risk factors for QT prolongation/arrhythmia (e.g., heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death in first-degree relatives <40 years);
7. Severe cardiovascular/cerebrovascular disease history；
8. History of other primary malignancies (except cured localized tumors like basal cell carcinoma, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate/cervix/breast, or subjects with other primary tumors showing no recurrence for ≥5 years);
9. Clinically confirmed active pneumonia at screening or history of interstitial lung disease;
10. Uncontrolled serous effusions requiring frequent drainage or medical intervention at screening (e.g., pleural/peritoneal/pericardial effusions needing additional intervention within 2 weeks after initial treatment, excluding cytological examination);
11. Brain metastases or spinal cord compression at screening (except those completing local therapy with ≥4-week steroid discontinuation and stable imaging/neurological symptoms for ≥4 weeks before treatment initiation);
12. Severe unhealed wounds/ulcers/fractures, or major surgery within 4 weeks before first dose, or planned elective surgery during study;
13. Clinically confirmed active HBV or HCV.Active HBV definition: HBcAb or HBsAg positive with HBV DNA above ULN; Active HCV definition: HCV antibody positive with HCV RNA above ULN;
14. Active tuberculosis confirmed clinically, or TP-Ab positive, or HIV-Ab positive, or history of immunodeficiency diseases/organ transplantation/allogeneic hematopoietic stem cell transplantation;
15. Significant bleeding tendency within 4 weeks before first dose, investigator-assessed high-risk of gastrointestinal hemorrhage/hemoptysis, or congenital bleeding disorders/coagulopathy;
16. Active infection requiring medication or unexplained fever ≥38.5°C during screening;
17. History of psychotropic substance abuse, alcoholism, or drug addiction;
18. Pregnancy or lactation at screening;
19. Persistent adverse reactions from prior antitumor therapy not recovered to CTCAE v5.0 ≤Grade 1 or baseline (except alopecia/nail changes/other investigator-deemed non-safety concerns);
20. Investigator-determined ineligibility for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
DLT（Phase 1a） | Up to approximately 21days
  Incidence rate and category of dose limiting toxicities (DLTs) during the first 21-day cycle of SYS6040 treatment
Frequency and severity of TEAE and SAE（Phase 1a） | Up to approximately 2years
  Assess safety and tolerability of SYS6040
RP2D (Phase 1a） | Up to approximately 2 years
  RP2D was determined based on the safety, tolerability, PK, immunogenicity data and efficacy information obtained
ORR（Phase 1b） | Up to approximately 2 years
  Objective response rate (ORR) as evaluated by Investigator (RECIST1.1).

SECONDARY OUTCOMES:
Peak time(Tmax)（phase 1a） | Up to approximately 2 years
  Peak time(Tmax) after a single administration of SYS6040
Maximum plasma concentration (Cmax) （phase 1a） | Up to approximately 2 years
  Cmax after a single administration of SYS6040
AUC 0-t（phase 1a） | Up to approximately 2 years
  Area under blood concentration - time curve(AUC 0-∞) after a single administration
AUC 0-∞（phase 1a） | Up to approximately 2 years
  Area under blood concentration - time curve(AUC 0-∞) after a single administration
Steady state peak concentration(Cmax,ss) （phase 1a） | Up to approximately 2 years
  Steady state peak concentration(Cmax,ss) after repeated administration
Steady state valley concentration(Cmin,ss) （phase 1a） | Up to approximately 2 years
  Steady state valley concentration(Cmin,ss) after repeated administration
DoR | Up to approximately 2 years
  Duration of response
DCR | Up to approximately 2 years
  Disease control rate
ORR（Phase 1a） | Up to approximately 2years
  Objective response rate (ORR) as evaluated by Investigator (RECIST1.1).
OS | Up to approximately 2 years
  Overall survival
PFS | Up to approximately 2 years
  Progression-free survival (PFS) as evaluated by Investigator (RECIST1.1).
Anti-SYS6040 antibodies | Up to approximately 2 years
  Anti-drug antibody (ADA) incidence and titer.
Adverse events (AEs)（Phase 1b） | Up to approximately 2 years
  Incidence and severity of AEs
Plasma concentrations of toxin-bound antibodies | Up to approximately 2 years
  Tests are conducted after administration of SYS6040.
Plasma concentrations of total antibodies | Up to approximately 2 years
  Tests are conducted after administration of SYS6040.
Plasma concentrations of free toxin | Up to approximately 2 years
  Tests are conducted after administration of SYS6040.

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchuan, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided